CLINICAL TRIAL: NCT01070121
Title: Treatment Efficacy and Toxicity in Rheumatoid Arthritis Database and Repository
Acronym: TETRAD
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Brigham and Women's Hospital (Other); Duke University (Other); Johns Hopkins University (Other); North Shore Medical Center (Other); Stanford University (Other); University of California, San Francisco (Other); University of Colorado, Denver (Other); University of Nebraska (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, S. Louis Bridges, MD, PhD, Director, Division of Clinical Immunology and Rheumatology, University of Alabama at Birmingham
Other Study IDs: F091007003
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; RA; Autoimmune Disease; Muscular Skeletal Disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, red blood cells, white blood cells, plasma, serum, DNA, RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RA patients/participants

SUMMARY:
To stimulate collaborative efforts of federal funding agencies, voluntary health agencies, professional organizations and industry partners to enable creation of a large, sustainable database and repository to better understand the molecular basis of treatment and rapidly accelerate translational research in RA.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is the most common inflammatory arthritis, affecting ~1% of the US population. Severity of RA varies from mild synovitis to joint destruction with associated disability and increased mortality. Methotrexate (MTX) is the major drug used to treat RA and the anchor drug for clinical trials of investigational new drugs (INDs) in RA. Eight biologic agents are currently FDA-approved for RA. No drug is effective in every patient, and there is great variability in toxicity and price.

The use of concomitant MTX and biologic agents has dramatically improved the outcomes of RA treatment in the US. This proposal is based on the premise the next major advance needed in the treatment of RA is not additional drugs, but rather a dramatic improvement in the efficiency and cost-effectiveness of the use of drugs for individual patients with RA. One of the hopes for modern medicine is the realization of "personalized" medicine, which allows accurate, quick prediction of which drug will be the most efficacious, least toxic, and least expensive for an individual patient.

One of the major obstacles to identifying clinically useful markers of treatment response in RA is the lack of cohorts with prospectively collected treatment response data coupled with biological samples. Because of the importance of this issue and the paucity of funding for such efforts, multiple efforts to establish single institution (using institutional funds) or multisite cohorts and repositories (typically dependent on private practitioners and pharmaceutical company support) are planned. To date, there has been no attempt to harmonize the efforts of the US academic RA research community to create a public resource.

Recognizing that building de novo cohorts within a short time frame is not feasible, our current proposal will fill a critical need: establishing an infrastructure of academic investigators to lay the foundation for future collaborative large-scale registries; and uniting the efforts of many organizations with the common goal of improving care of RA patients. This project will facilitate future research that will result in significant, publicly visible improvements in health care. Identifying predictors of treatment response in RA will lead to rapid, early institution of optimal drugs rather than a "hit or miss" sequential approach; reduce adverse events; improve patient compliance; and lead to substantial reduction in the cost of health care. By unifying the efforts of academic researchers, we can create unique resources, such as a bank of cryopreserved blood cells to allow sophisticated immunologic research to dissect molecular signals of successful treatment of RA.

In order to determine the feasibility of this infrastructure for prospectively collecting data and samples we will enroll a small number of participants (10/site/year for each of 2 years, for a total of 200 participants).

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 years or older;
2. Diagnosis of RA based on the cumulative presence of at least 4 of 7 ACR Criteria;
3. Willing and able to provide informed consent; and

One of the following:

* Starting MTX OR
* Previous or current use of Methotrexate and starting (or switching to) any of the following medications (with or without MTX)

  * Etanercept
  * Infliximab
  * Adalimumab
  * Rituximab
  * Abatacept
  * Golimumab
  * Certolizumab
  * Tocilizumab

There is no minimum disease activity (number of swollen joints, DAS28, CRP or ESR, etc.) necessary for enrollment. Treatment decisions are entirely at the discretion of the treating rheumatologist.

There are no combinations of drugs to be excluded, except those that do not include at least one of the seven drugs noted above.

Use of corticosteroids (oral, parenteral, intra-articular) is allowed, but must be recorded.

Exclusion Criteria:

Concomitant diagnosis of RA and systemic lupus erythematosus, juvenile arthritis, psoriatic arthritis, hepatitis C infection, current pregnancy or lactation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Speciality/referral clinic, Community
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The number of enrolled patients will be used as a measure of success. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: S. Louis Bridges, Jr., MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - University of Colorado in Denver, Aurora, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - North Shore Medical Center (LIJ Health System), Lake Success, New York
  - Duke University, Durham, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Ormseth MJ, Yancey PG, Solus JF, Bridges SL Jr, Curtis JR, Linton MF, Fazio S, Davies SS, Roberts LJ 2nd, Vickers KC, Kon V, Michael Stein C; TETRAD Investigators. Effect of Drug Therapy on Net Cholesterol Efflux Capacity of High-Density Lipoprotein-Enriched Serum in Rheumatoid Arthritis. Arthritis Rheumatol. 2016 Sep;68(9):2099-105. doi: 10.1002/art.39675. PMID 26991245